CLINICAL TRIAL: NCT04745390
Title: A Phase III Randomized Trial of Standard Dose Stereotactic Body Radiation Therapy (SBRT) Versus Radiobiologically-Guided Dose Selected SBRT in Primary or Secondary Liver Carcinoma (SAVIOR).
Brief Title: Standard Versus Radiobiologically-Guided Dose Selected SBRT in Liver Cancer
Acronym: SAVIOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Lock, Radiation Oncologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAVIOR
Record Dates: First submitted 2021-01-23; First posted 2021-02-09 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma; Liver Metastases
Keywords: Hepatocellular Carcinoma; Radiation Therapy; Stereotactic Body Radiation Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Dose Radiation (Active Comparator): Patients in the standard arm will receive a standard dose of 2000cGy in 5 fractions using simple CT planning. IMRT is allowed. Treatment will be every second day excluding weekends and holidays.
  Interventions: Radiation: Radiation therapy
- Personalized Dose Selection Radiation (Experimental): Patients in the experimental arm will receive individually selected prescription dose guided by radiobiological parameters described below, preferably delivered in 5 fractions every other day, excluding weekends and holidays. Volumetric-modulated arc therapy (VMAT) is the preferred planning technique. Typical planning uses 2 arcs, <=10MV and FFF mode where possible as almost all liver treatments are gated). In the event of multiple lesions, multiple isocentres are allowed. Often lateral isocentre shifts are significant and therefore arc ranges should be chosen to minimize collision risk. Treatment will be every second day excluding weekends and holidays.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Patients will be randomized between standard of care palliative irradiation of 2000cGy in 5 fractions (Arm 1) versus radiobiologically guided dose selection also in 5 fractions (Arm 2). For all patients randomized, radiation is to be delivered in 5 fractions delivered over 5 to 15 days.

SUMMARY:
Radiation is a standard treatment option for patients with liver cancer. Unfortunately, the tumour grows after radiation in many patients and radiation can harm normal tissues. A new treatment using a specialized radiation procedure called Stereotactic body radiotherapy (SBRT) may increase the chance to control liver cancer and reduce the chance of harm to normal tissues. SBRT allows radiation treatments to be focused more precisely, and be delivered more accurately than with older treatments. SBRT has become a routine treatment. Further research has found that specialized computer programs can possibly guide the selection of an appropriate SBRT dose. This is called radiobiological guidance. However, this has not yet been proven to improve outcomes and/or reduce toxicity.

Therefore, the purpose of this study is to find out if SBRT at standard dose versus SBRT guided by radiobiological techniques is better for you and your liver cancer.

DETAILED DESCRIPTION:
Primary and secondary (aka liver metastases) hepatobiliary cancer cause substantial morbidity in an increasing number of patients primarily due to the fact that only a minority of patients are suitable for curative treatment; a majority of patients have limited options and have dismal survival rates. First, primary cancers of the hepatobiliary tract are one of the most common malignancies internationally. Though they occur less frequently in the industrialized world; however, the incidence of primary hepotobiliary cancer is one of the fastest rising cancers in North America. Treatments for unresectable hepatobiliary cancer, including chemotherapy and hepatic arterial embolization are associated with low response rates and very poor survival. Second, metastatic disease to the liver is common and, like primary hepatobiliary cancer, causes significant morbidity and mortality. Metastatic colorectal cancer to the liver is a common pattern of spread, sometimes as the only site of metastatic disease. Autopsy studies have shown that 40% of colon cancer patients fail with disease confined to the liver. Approximately 50% of metastatic deaths from breast and prostate cancers are associated with liver metastases: 43,000 women and 34,000 men per year. This has led to the hypothesis that not all metastases are diffuse and that "oligometastasis" can occur where aggressive local therapy to the oligometastasis may lead to long-term control of disease. This hypothesis is gaining support over the currently held belief that metastases are always systemic. Evidence for the oligometastasis theory is found in surgical series of treated oligometastases of the colon, sarcoma, melanoma and breast. If metastases were truly confined to the liver, and if effective therapy for the localized intrahepatic disease existed, aggressive local therapy may lead to cure in some patients. Given that patients with liver lesions (both primary and secondary) currently have few options, the potential gains in national cancer survival are substantial if an effective high-dose focal liver radiation treatment regimen could be delivered safely and effectively.

Recent technological advances have made it possible to deliver high doses of radiation therapy precisely to small tumours while preserving function in critical structures surrounding the lesion. With these techniques, control rates in excess of 80% have been achieved in patients with metastasis from lung, breast, renal, and other cancers. We hypothesize that similar control rates may be feasible using stereotactic radiotherapy for liver cancers.

External beam radiotherapy has long been considered to have a very limited role in the treatment of liver tumours. This has historically been because minimum dose required for local ablation exceeded the dose that would result in liver toxicity which can be morbid and cause death. The technical development of stereotactic body radiation therapy (SBRT) renewed interest in radiation for HCC. For SBRT, advanced techniques are used to very accurately deliver a high total dose to the target in a small number of daily fractions while avoiding dose delivery to surrounding healthy structures. This research in HCC was done mainly by two groups, in Michigan and Stockholm, who demonstrated that the delivery of high doses of radiation to limited volumes of the liver had promising results in terms of local control and survival with acceptable toxicity. SBRT is offered as an ablative radical local treatment as opposed to low palliative doses. In total as of 2015, eleven primary series reported on tumour response and survival of around 300 patients who have been treated with stereotactic body radiation therapy as primary therapy for HCC. The reported percentage of objective responses defined as complete and partial was ≥64% in 7 of 8 series. Median survival between 11.7 and 32 months has been observed. Toxicity, based on multiple case series trials, indicate that the treatment is considered safe. The most common CTC grade 3-4 toxicity was elevation of liver enzymes.

However, there is no accepted dose or dose regimen. The reason for a lack of liver SBRT's acceptance into practice is this lack of a standard regimen and the fact that most dose selection studies are based on anecdotal experience or small single institution dose escalation studies. Furthermore, known risks of harm, including death, have been shown in dose escalation studies. Given the relative heterogeneity of liver cancer patients, small sample sizes and high risk of harm, a consensus dose regimen that can be tested remains elusive.

One solution is to individualize dose selection to decrease the impact of heterogeneity of patient anatomy, type of cancer, size of lesion and motion. The liver tolerance to external beam irradiation depends on the volume treated and the fractionation schedule. Lawrence, et al found that patients who developed grade III or IV radiation induced liver disease (RILD) tended to receive a higher mean dose and have less sparing of normal liver than those who did not. In the original analysis, none of the 45 patients who received a mean dose to the whole liver of less than 37 Gy (in 1.5 Gy per fraction bid) developed RILD, while 9 of 34 patients who received a mean dose of more than 37 Gy developed this complication. Another study from the University of Michigan looked at 26 patients with hepatobiliary cancer treated with radiation doses up to 72.6 Gy, in 1.5 Gy bid and concurrent intrahepatic fluorodeoxyuridine administration. Patients treated with a component of 36 Gy whole liver radiation were more likely to develop RILD compared to those treated with focal high-dose radiation with no whole liver radiation. These studies indicate that by using modern conformal radiation planning it is possible to deliver tumouricidal doses of radiation safely. More recently, we have developed a better understanding of the relationship between dose, volume of liver irradiated and RILD, based on an analysis of over 200 patients with hepatic malignancies treated at the University of Michigan. This analysis demonstrates that for a small effective liver volume irradiated, far higher doses of radiation can be prescribed than previously estimated. In addition to the dose and volume irradiated, several other factors were significantly associated with increased the risk of RILD, including use of BUdR chemotherapy (versus FuDR), primary hepatobiliary cancer diagnosis (versus metastatic cancer diagnosis) and male sex. Excluding 32 patients treated with BudR, leaving 169 patients treated with 1.5 Gy bid with concurrent FudR, the mean liver dose associated with a 5% risk of RILD for patients with metastases and primary hepatobiliary cancer were 37 Gy and 32 Gy, in 1.5 Gy bid. Assuming an alpha/beta ratio for the liver of 2.5 Gy, the corresponding mean liver doses associated with a 5% risk of RILD are 33 Gy and 28 Gy in 2 Gy per fraction, and 28.2 Gy and 25.1 Gy in 10 fractions, for metastases and primary liver cancer respectively. This radiobiological guidance has been used at the London Regional Cancer Program since 2004 with a REB approved, prospectively collected case series. This radiobiologically-guided individualized dose selection is now used routinely in London, has shown a very good tolerability and can be implemented immediately. Doses can be escalated and de-escalated to account for variation in patient anatomy, tumour and normal tissue motion, comorbidities, size of lesion, number of lesions and function of the normal liver. However, the value of this new technique relative to palliative treatment is unknown. In particular, is there a survival advantage to dose escalation based on the oligometastases theory.

For unresectable cases, SBRT has been shown to be a safe alternative for patients with few, if any, options. However, neither the appropriate dose regimen nor impact on important clinical endpoints, including survival has been determined; and no randomized trials have been published to guide management. Individualized dose selection based on radiobiological parameters promises a safe dose escalation or de-escalation for each patient. Therefore, a phase III randomized clinical study comparing palliative external beam radiation and a radiobiologically

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients include patients with any of the following:

   * Primary hepatobiliary cancer confirmed pathologically or,
   * Non-lymphoma liver metastases confirmed pathologically or,
   * Radiographic liver lesions most consistent with metastases, in a patient with known pathologically proven non-lymphoma cancer and a previously negative CT or MRI of the liver or,
   * Hepatocellular carcinoma diagnosed with vascular enhancement of the lesion consistent with hepatocellular carcinoma, and with an elevated AFP, in the setting of cirrhosis or chronic hepatitis.
2. ≤ 5 liver lesions measurable on a contrast-enhanced liver CT or MRI performed within 90 days prior to study entry.
3. Primary liver lesion or liver metastases measuring ≤ 25 cm.
4. Extrahepatic cancer is permitted if liver involvement is judged to be life-limiting
5. No contraindications to radiotherapy
6. Patient must be judged medically or surgically unresectable
7. Zubrod Performance Scale = 0-3
8. Age > 18
9. Systemic treatment including multikinase inhibitors and immunotherapy are allowed.

   Multikinase inhibitors must be held 2 weeks prior to radiation and may be restarted 1 week post radiation.
10. Previous liver resection or ablative therapy is permitted
11. Chemotherapy must be completed at least 2 weeks prior to radiation therapy and not planned to be administered for at least 1 week (for anthracyclines at least 4 weeks) after completion of treatment.
12. Life expectancy > 6 months.
13. Women of childbearing potential and male participants must practice adequate contraception.

Exclusion Criteria:

1. Severe cirrhosis or liver failure defined as Child Pugh >B7
2. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
3. Severe, active co-morbidity, defined as limiting the patient's life to less than 6 months
4. Active hepatitis or clinically significant liver failure. Treated hepatitis is permitted.
5. Pregnancy, nursing women, or women of childbearing potential, and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6 months
  What will be overall survival of patients in two arms? How many patients progressed in each arm after receiving radiation?
Treated lesion progression | 6 months
  What is the local radiated lesion progression rate?

SECONDARY OUTCOMES:
Response rate - Modified RECIST criteria | 6 months
  To calculate the response rate for each patient according to the modified RECIST criteria.
  * Complete Response: Disappearance of all target lesions
  * Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD
  * Progressive Disease: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Extrahepatic failure | From date of randomization until the date of first documented extrahepatic failure or date of death from any cause, whichever came first, assessed up to 2 years
  Number of patients presented with Extrahepatic failure which defined by Any new lesion present outside of the liver organ.
Time to intrahepatic progression | From date of randomization until the date of first documented intrahepatic progression or date of death from any cause, whichever came first, assessed up to 2 years
  To calculate the time in months or years for cancer recurrence after treatment.
Toxicity from the intervention | 6 months
  Evaluate acute and long-term G3 or larger toxicity based on NCI-CTCAE 5.0 score system. Grade 1 to Grade 5. Higher the grade more severe is the toxicity.
Comparison of Quality of Life (QOL) Using a Standardly-Used Validated Instrument. Specifically, measures of physical, social/family, and functional well being. Overall symptoms, function, global health status will also be compared. | Pre-treatment, weekly during treatment, 1 month post treatment, 3 month post treatment, every 3 months up to 5 years.
  EORTC QLQ-C30(European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) comprises 5 functional, 3 symptom, 6 single symptom and 1 global health status scale. A higher score denotes a better quality of life for the function and global health scales. A lower score on the symptom and single item scales indicates a lower state of the patient. Overall score will be the primary measure. Scale is 0-100 points.
Comparison of Quality of Life (QOL) Using a Standardly-Used Validated Instrument. Specifically, measures of physical, social/family, and functional well being. Overall symptoms, function, global health status will also be compared. | Pre-treatment, weekly during treatment, 1 month post treatment, 3 month post treatment, every 3 months up to 5 years.
  FACT-Hep(Functional Assessment of Cancer Therapy-Hepatobiliary questionnaire) is a specific to liver patient quality of life instrument assessing the functional quality of life of patients with hepatobiliary cancer. It has 45 Likert-type items with well-being domains of physical, social/family, emotional, functional plus a hepatobiliary cancer subscale. Aggregate overall lower scores denote a better state of the patient (leading some items to be reverse scored). Overall score will be the primary measure. Scale is 0-180 points.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lock, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghouri YA, Mian I, Rowe JH. Review of hepatocellular carcinoma: Epidemiology, etiology, and carcinogenesis. J Carcinog. 2017 May 29;16:1. doi: 10.4103/jcar.JCar_9_16. eCollection 2017. PMID 28694740
- [Background] De P, Dryer D, Otterstatter MC, Semenciw R. Canadian trends in liver cancer: a brief clinical and epidemiologic overview. Curr Oncol. 2013 Feb;20(1):e40-3. doi: 10.3747/co.20.1190. PMID 23443230
- [Background] Jarnagin W, Chapman WC, Curley S, D'Angelica M, Rosen C, Dixon E, Nagorney D; American Hepato-Pancreato-Biliary Association; Society of Surgical Oncology; Society for Surgery of the Alimentary Tract. Surgical treatment of hepatocellular carcinoma: expert consensus statement. HPB (Oxford). 2010 Jun;12(5):302-10. doi: 10.1111/j.1477-2574.2010.00182.x. PMID 20590903
- [Background] Klein J, Dawson LA. Hepatocellular carcinoma radiation therapy: review of evidence and future opportunities. Int J Radiat Oncol Biol Phys. 2013 Sep 1;87(1):22-32. doi: 10.1016/j.ijrobp.2012.08.043. Epub 2012 Dec 6. PMID 23219567
- [Background] Mazzaferro V, Regalia E, Doci R, Andreola S, Pulvirenti A, Bozzetti F, Montalto F, Ammatuna M, Morabito A, Gennari L. Liver transplantation for the treatment of small hepatocellular carcinomas in patients with cirrhosis. N Engl J Med. 1996 Mar 14;334(11):693-9. doi: 10.1056/NEJM199603143341104. PMID 8594428
- [Background] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Background] Shim SJ, Seong J, Han KH, Chon CY, Suh CO, Lee JT. Local radiotherapy as a complement to incomplete transcatheter arterial chemoembolization in locally advanced hepatocellular carcinoma. Liver Int. 2005 Dec;25(6):1189-96. doi: 10.1111/j.1478-3231.2005.01170.x. PMID 16343071
- [Background] Borgelt BB, Gelber R, Brady LW, Griffin T, Hendrickson FR. The palliation of hepatic metastases: results of the Radiation Therapy Oncology Group pilot study. Int J Radiat Oncol Biol Phys. 1981 May;7(5):587-91. doi: 10.1016/0360-3016(81)90370-9. No abstract available. PMID 6168623
- [Background] Emami B, Lyman J, Brown A, Coia L, Goitein M, Munzenrider JE, Shank B, Solin LJ, Wesson M. Tolerance of normal tissue to therapeutic irradiation. Int J Radiat Oncol Biol Phys. 1991 May 15;21(1):109-22. doi: 10.1016/0360-3016(91)90171-y. PMID 2032882
- [Background] Lax I, Blomgren H, Naslund I, Svanstrom R. Stereotactic radiotherapy of malignancies in the abdomen. Methodological aspects. Acta Oncol. 1994;33(6):677-83. doi: 10.3109/02841869409121782. PMID 7946448
- [Background] McGinn CJ, Ten Haken RK, Ensminger WD, Walker S, Wang S, Lawrence TS. Treatment of intrahepatic cancers with radiation doses based on a normal tissue complication probability model. J Clin Oncol. 1998 Jun;16(6):2246-52. doi: 10.1200/JCO.1998.16.6.2246. PMID 9626227
- [Background] Dawson LA, McGinn CJ, Normolle D, Ten Haken RK, Walker S, Ensminger W, Lawrence TS. Escalated focal liver radiation and concurrent hepatic artery fluorodeoxyuridine for unresectable intrahepatic malignancies. J Clin Oncol. 2000 Jun;18(11):2210-8. doi: 10.1200/JCO.2000.18.11.2210. PMID 10829040
- [Background] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075
- [Background] Cardenes HR, Price TR, Perkins SM, Maluccio M, Kwo P, Breen TE, Henderson MA, Schefter TE, Tudor K, Deluca J, Johnstone PA. Phase I feasibility trial of stereotactic body radiation therapy for primary hepatocellular carcinoma. Clin Transl Oncol. 2010 Mar;12(3):218-25. doi: 10.1007/s12094-010-0492-x. PMID 20231127
- [Background] Mendez Romero A, Wunderink W, Hussain SM, De Pooter JA, Heijmen BJ, Nowak PC, Nuyttens JJ, Brandwijk RP, Verhoef C, Ijzermans JN, Levendag PC. Stereotactic body radiation therapy for primary and metastatic liver tumors: A single institution phase i-ii study. Acta Oncol. 2006;45(7):831-7. doi: 10.1080/02841860600897934. PMID 16982547
- [Background] Tse RV, Hawkins M, Lockwood G, Kim JJ, Cummings B, Knox J, Sherman M, Dawson LA. Phase I study of individualized stereotactic body radiotherapy for hepatocellular carcinoma and intrahepatic cholangiocarcinoma. J Clin Oncol. 2008 Feb 1;26(4):657-64. doi: 10.1200/JCO.2007.14.3529. Epub 2008 Jan 2. PMID 18172187